CLINICAL TRIAL: NCT01211613
Title: A Comparison of Chiropractic Manipulation Methods and Standard Medical Care for Low Back Pain
Brief Title: Chiropractic Manipulation and Medical Care for Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Michael Schneider, DC, PhD, DC, PhD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO10040327; 4R00AT004196-03 (NIH)
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Low Back Pain
Keywords: Manipulation; Chiropractic; Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Manual Manipulation (Experimental): Doctor of chiropractic will apply manual high-velocity low-amplitude thrust to lumbar spine of research participants.
  Interventions: Procedure: Manual Manipulation
- Mechanical Manipulation (Experimental): Doctor of chiropractic will apply a mechanically-assisted thrust to the lumbar spine of research participants using the Activator IV Instrument.
  Interventions: Device: Mechanically-assisted manipulation
- Standard Medical Care (Active Comparator): Patients will receive an examination with a physician who is board certified in physical medicine and rehabilitation. Treatment will consist of medical monitoring of the patient's condition over 4 weeks (baseline and 2 follow up exams) and a prescription for over-the-counter anti-inflammatory medications if indicated.
  Interventions: Other: Standard Medical Care

INTERVENTIONS:
Procedure: Manual Manipulation — Doctor of chiropractic will apply manual high-velocity low-amplitude thrust to lumbar spine of research participants.
  Arms: Manual Manipulation
Device: Mechanically-assisted manipulation — Doctor of chiropractic will use the Activator Instrument to apply a mechanically-assisted thrust to the lumbar spine of research participants.
  Other Names: Activator IV Instrument: FDA approval# K003185
  Arms: Mechanical Manipulation
Other: Standard Medical Care — Patients will receive an examination with a physician who is board certified in physical medicine and rehabilitation. Treatment will consist of medical monitoring of the patient's condition over 4 weeks (baseline and 2 follow up exams) and a prescription for over-the-counter anti-inflammatory medications if indicated.
  Arms: Standard Medical Care

SUMMARY:
The investigators will be comparing the effectiveness of two types of chiropractic manipulation and standard medical care for patients with a recent onset of low back pain. The two types of chiropractic treatments being compared will be hands-on (manual) manipulation and mechanical-assisted (Activator) manipulation. The standard medical care will consist of a medical examination and prescription for over-the-counter anti-inflammatory medication.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years of age
* Ability to read and write English
* Experiencing a new episode of low back pain (LBP) with onset in the past 3 months
* Oswestry Disability Index score between 20-70 points (0-100 scale)
* Numeric pain rating score between 3-8 points (0-10 scale)

Exclusion Criteria:

* Prior history of lumbar spine surgery
* History of unstable spondylolisthesis, spinal stenosis, or scoliosis > 20°
* Signs or symptoms suggestive of nerve root tension and/or neurological deficit in the lower extremity
* History of metastatic cancer, osteoporosis, long-term corticosteroid use, or any other red flags of serious illness including the following: unexplained weight loss of >10% of body weight, spinal pain associated with fever, and severe night pain unrelieved by medication
* Receiving any physical therapy, chiropractic therapy, or any other manual therapy for this episode of LBP (within the past 3 months)
* Receiving any on-going medical care for this episode of low back pain
* Current use of opiate or other prescription medications for low back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2010-11; Primary Completion 2013-03 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Schneider, PhD, DC, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center: Center for Integrative Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Schneider MJ, Brach J, Irrgang JJ, Abbott KV, Wisniewski SR, Delitto A. Mechanical vs manual manipulation for low back pain: an observational cohort study. J Manipulative Physiol Ther. 2010 Mar-Apr;33(3):193-200. doi: 10.1016/j.jmpt.2010.01.010. PMID 20350672
- [Derived] Tonelli Enrico V, Schneider M, Haas M, Vo N, Huang W, McFarland C, Weber N, Sowa G. The association of biomarkers with pain and function in acute and subacute low back pain: a secondary analysis of an RCT. BMC Musculoskelet Disord. 2022 Dec 5;23(1):1059. doi: 10.1186/s12891-022-06027-9. PMID 36471334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 112 patients with a new episode of low back pain from the general population of the Greater Pittsburgh Metropolitan region. Recruitment took place during the period of time between November 2010 and April 2013.
Pre-assignment Details: 197 patients were screened for potential eligibility. We excluded 85 patients for not meeting the inclusion criteria. Of the 40 patients randomized to Standard Medical Care, 3 never showed up for their first visit and 2 were withdrawn by the PI before receiving any treatments; leaving only 35 in that arm.
Period: Overall Study
Arm/Group | Manual Manipulation | Mechanical Manipulation | Standard Medical Care
Started | 37 | 35 | 35
Completed | 34 | 33 | 33
Not Completed | 3 | 2 | 2
Not completed — Lost to Follow-up | 2 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Manipulation | Mechanical Manipulation | Standard Medical Care | Total
Number analyzed (Participants) | 37 | 35 | 35 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (15.3) | 40.4 (28.8) | 41.3 (27.4) | 41.1 (28.8)
Gender [Count of Participants; unit: Participants]
  Female | 25 | 21 | 21 | 67
  Male | 12 | 14 | 14 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 9 | 11 | 29
  White | 23 | 22 | 22 | 67
  More than one race | 3 | 4 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Oswestry Low Back Pain Disability Index
Description: The Oswestry (OSW) Questionnaire provides the level of self-reported impairment of activity of daily living (ADLs) due to low back pain. There are 10 items in the OSW, each rated on a Likert scale from 0-5. The total range of possible scores is from 0 -50, which is converted to a percentage ranging from 0-100. The percentage of self-reported disability ranges from 0='no impairment' to 100='complete impairment'. Our statistical analysis looked at the change in OSW score (in percentage points) from baseline to 4 weeks (post treatment).
Time Frame: 4 weeks (post treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Manual Manipulation | Mechanical Manipulation | Standard Medical Care
Number analyzed (Participants) | 37 | 35 | 35
units on a scale | -16.0 (14.1) | -8.9 (11.9) | -9.5 (14.4)
Statistical Analysis 1: Comparison: Manual Manipulation vs Mechanical Manipulation vs Standard Medical Care; Test type: Superiority or Other; p = 0.009, Regression, Linear — The p value above relates to the comparison of differences in baseline/4-week Oswestry change scores between manual and mechanical manipulation methods (primary hypothesis). A priori threshold for statistical significance was set at p < 0.05; Linear regression model was adjusted for these covariates: baseline Oswestry score, age, and treatment expectancy; Mean Difference (Final Values) = 10, Standard Deviation 14

2. Secondary Outcome: Numeric Pain Rating Score.
Description: Self-reported level of low back pain. We used the mean of 3 numeric pain rating scales: 1) current pain; 2) worst pain in the past 24 hours; and 3) average pain over the past week. Three individual 0 to 10 Likert scales were anchored by 0 indicating "no pain" and 10 indicating "unbearable pain". Our primary statistical analysis looked at the change in pain scores from baseline to 4 weeks (post treatment).
Time Frame: 4 weeks (post treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Manual Manipulation | Mechanical Manipulation | Standard Medical Care
Number analyzed (Participants) | 37 | 35 | 35
units on a scale | -3.7 (1.5) | -2.6 (1.6) | -1.9 (2.2)
Statistical Analysis 1: Comparison: Manual Manipulation vs Mechanical Manipulation vs Standard Medical Care; Test type: Superiority or Other; p = 0.002, Regression, Linear — The p value above relates to the comparison of differences in baseline/4-week Numeric pain change scores between manual and mechanical manipulation methods (secondary hypothesis). A priori threshold for statistical significance was set at p < 0.05; Linear regression model was adjusted for these covariates: baseline Numeric pain score, age, and treatment expectancy

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at each treatment visit in each of the 3 treatment arms, over the course of the entire 4-week treatment period.
Arm/Group | Manual Manipulation | Mechanical Manipulation | Standard Medical Care
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/37 | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes